CLINICAL TRIAL: NCT04035408
Title: Tracking the Natural History of Facial Skin Health in Pre and Peri Menopausal Breast Cancer Patients Undergoing Chemotherapy and / or Endocrine Therapies: A Feasibility Study
Brief Title: Facial Skin Health Tracking Feasibility in Breast Cancer Patients
Status: Withdrawn | Type: Observational
Why Stopped: Low/No Accrual
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 18-2444.cc
Record Dates: First submitted 2019-07-10; First posted 2019-07-29 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Breast Cancer Female

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All subjects: All the enrolled subjects will be considered for the assessment of the primary and secondary outcomes.
  Interventions: Other: Skin health assessment

INTERVENTIONS:
Other: Skin health assessment — Assess and measure the natural history of facial skin changes in pre and perimenopausal women undergoing chemotherapy and/or endocrine therapy for breast cancer

SUMMARY:
This feasibility study will assess if tracking objective and subjective facial skin changes over time is acceptable to pre and perimenopausal women undergoing chemotherapy and/or endocrine therapy for breast cancer. There is no intervention arm and no control group. Skin health will be assessed through the instruments described below, and subjective data will be collected with self-administered questionnaires.

DETAILED DESCRIPTION:
There are no studies objectively assessing changes to facial skin health in this population, but tools exist to objectively measure changes thus we have chosen to use those tools to measure skin health. Before embarking on an intervention study showing improvement in skin health and patients' self-image and QOL, we first need to see if 1) it is feasible to measure changes in skin health in this population and 2) if skin health does objectively change over the course of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form
2. Stated willingness to comply with all study procedures and be available for the duration of the study
3. Be a pre or perimenopausal woman age 18 or over
4. Be a patient with a new diagnosis of breast cancer who plans to undergo systemic chemotherapy or endocrine therapy, but who has not yet started treatment

Exclusion Criteria:

1. Postmenopausal status (one year without a menstrual period)
2. Pregnant women (pregnancy test not required)
3. Prior cancer diagnosis of any type other than breast cancer
4. History of prior treatment with chemotherapy or radiation therapy
5. Chronic skin disease including scleroderma, discoid lupus, atopic dermatitis, rosacea, eczema, or psoriasis
6. Use of a retinoid-based prescription facial skin product within the past 11 month

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — pre or perimenopausal woman age 18 or over
Study Population: Our baseline skin health self-assessment tool accounts for smoking status, sun exposure, and sunscreen use and this will factor into our assessments/comparison to age and ethnicity matched norms. Sun exposure will likely affect skin age differences at baseline but should not affect the skin aging over the duration of the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Percentage of compliance in each of the 4 assessment tools | 3 years
  defined as the percentage of patients completing all the scheduled assessments under each assessment tool. The percentage of compliance will be summarized and the associated 90% confidence interval reported. If the percentage of compliance is 80% or higher under each assessment tool, the study will be considered feasible.

SECONDARY OUTCOMES:
Changes in skin health over the duration of the study (4 assessment points) | 3 years
  Difference in skin health at each assessment from baseline will be calculated which will be divided by the standard deviation of the difference to obtain the effect size of the change at each assessment time post baseline
Changes in body image / skin QOL at end of treatment compared to baseline | 3 years
  Skindex16 will be used to assess. Skin traits will be rated from 0 (never bothered) to 6 (always bothered). The max score being 96, the least being 0.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No